CLINICAL TRIAL: NCT04822454
Title: Early Exposure of Medical Students to Night Shifts: Impact on Well-being and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, Anthony Kerbage, Principal Investigator, PGY-1 Resident of Internal Medicine, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: StJosephBeirut
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Medical Students Well-being and Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Night shift shadowing program (Experimental): Medical students who participated in a night shift shadowing program prior to their first official night shifts
  Interventions: Other: Night shift shadowing program
- No night shift shadowing program (No Intervention): Medical students who did not participate in the night shift shadowing program prior to their first official night shifts

INTERVENTIONS:
Other: Night shift shadowing program — Our population, made up of 70 students, was divided into two randomly randomized groups: 31 (44.3%) had five night shift shadowing duty prior to their first official night shifts, and 39 (55.7%) did not participate in the shadowing program.
  Arms: Night shift shadowing program

SUMMARY:
This is an interventional study assessing the impact of 'shadowing night shifts' early during medical school, on the wellbeing and level of anxiety of a students during their first official night shifts.

ELIGIBILITY:
Inclusion Criteria:

* Students of the class of 2021 at the Faculty of Medicine of Saint Joseph University in their fifth year (Med 2).

Exclusion Criteria:

* student who has already been on call during internships in Lebanon or abroad, as well as students in other medical years.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 6 months
  After the shadowing program is completed, both groups of medical students (those who participated in the shadowing program and those who did not), have to fill a questionnaire that assesses their wellbeing and level of anxiety regarding their first official night shifts. Our primary outcome is to evaluate the impact of the shadowing program on medical students well-being and their level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, N/A (n/a), Lebanon

IPD SHARING:
Plan to Share IPD: Undecided